CLINICAL TRIAL: NCT03476473
Title: Early Detection of Respiratory Disorders in Psychosis
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Fundación Marques de Valdecilla (Other)
Collaborators: Instituto de Investigación Marqués de Valdecilla (Other); Consorcio Centro de Investigación Biomédica en Red (CIBER) (Other Government)
Responsible Party: Principal Investigator, Benedicto Crespo-Facorro, Associate Professor of Psychiatry, Fundación Marques de Valdecilla
Other Study IDs: RESP_10PAFIP
Record Dates: First submitted 2018-03-19; First posted 2018-03-26 (Actual); Last update posted 2020-12-16 (Actual); Status verified 2020-12

CONDITIONS: Schizophrenia; Psychosis; Chronic Respiratory Disease
Keywords: Asthma; Chronic obstructive pulmonary disease; Spirometry; Lung disease; Smoke
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders; Asthma; Pulmonary Disease, Chronic Obstructive; Lung Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aims to evaluate the presence of lung function impairment in a sample of patients diagnosed with non-affective psychosis.

DETAILED DESCRIPTION:
Asthma and chronic obstructive pulmonary disease (COPD) are chronic respiratory disorders with high prevalence in the general population. Tobacco smoking is the leading risk factor for COPD, and has been associated with higher risk for uncontrolled asthma. Tobacco smoking is widely extended in the general population and is highly associated with cannabis use, which is the most consumed illicit drug in Spain. Other described risk factors for poor lung function are metabolic alterations such as insulin resistance and diabetes, and even abdominal obesity. Patients with psychosis present remarkably higher prevalence of tobacco and cannabis consumption than the general population and higher risk for developing metabolic alterations such as obesity and diabetes at the long-run.

Despite these premises, the effect of metabolic alterations and tobacco and cannabis smoking on the respiratory health has been poorly studied. Previous studies, mainly based on patients' registers showed an increased risk for COPD and uncontrolled asthma in patients with psychosis. Few studies have analysed this relation using lung function tests (spirometry), reporting reduced spirometry values in patients with schizophrenia compared with healthy controls. But little data is available on the possible causative relation of smoking (tobacco and cannabis) and metabolic alterations of COPD and un-controlled asthma in psychosis.

Based on the available scientific evidence, the investigators hypothesize that patients with psychosis will present differences in prevalence and severity of lung disease and poorer lung function, compared with the general (non-psychiatric) population, probably related to smoking (tobacco and cannabis) and metabolic alterations.

The research project would be implemented as part of a larger prospective longitudinal study on first episode non-affective psychosis, in the First Episode Psychosis Clinical Program (PAFIP). In particular, the project would be part of the "10 PAFIP study", in which those patients that had been included in the PAFIP program 10 years ago will be extensively evaluated (e.g.: clinical, neuroimaging, neuro-psychological, and metabolic evaluations) in order to analyse the long-term progress of the psychosis.

Regarding the present project, a respiratory health status evaluation would be carried out cross-sectionally at this time-point (after 10 years of initiated the psychotic illness). Lung health status would be evaluated through functional test using spirometer. The clinical respiratory status would be evaluated using the following scales: the COPD Assessment Test (CAT) and the modified Medical Research Council (mMRC) Questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Patients followed in the First Episode Psychosis Clinical Program (PAFIP) from February 2001 to December 2007.
* Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition (DSM-IV) criteria of brief psychotic disorder, schizophreniform disorder, schizophrenia or schizoaffective disorder.

Exclusion Criteria:

* Meeting DSM-IV criteria for drug dependence.
* Meeting DSM-IV criteria for mental retardation.
* Having a history of neurological disease or head injury.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Individuals included in the Longitudinal Long-term Study of First Episode Psychosis Clinical Program (10 PAFIP) at the University Hospital Marqués de Valdecilla (Santander - Cantabria).
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2018-02-16 (Actual); Primary Completion 2018-03-26 (Actual); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
The incidence of COPD and asthma diagnosed by spirometry. | 10 years
  The spirometer variables will be forced vital capacity (FVC) (i.e. the maximal volume of air, in litres, that can be forcefully expelled from the lungs after maximal inhalation) and forced expiratory volume in 1 s (FEV1) (i.e. the volume of air that can be forcefully expelled from the lungs in the first second after maximal inhalation, in litres). From a minimum of two technically acceptable and consistent efforts, the highest readings of FEV1 and FVC will be recorded and used in the analyses. Spanish reference values will be used to compute the individual FEV1 and FVC values as a percentage of those predicted for corresponding age, gender and height in healthy, non-smoking adults. Based on spirometry results, pulmonary obstruction is defined as a FEV1/FVC <70%; and restriction as a FVC <80% of the predicted value and a FEV1/FVC >70% to exclude obstruction.

CONTACTS AND LOCATIONS:
Overall Officials: Ana Viejo Casas, Principal Investigator — Instituto de Investigación Marqués de Valdecilla
Locations (1):
- University Hospital Marqués de Valdecilla, Santander, Cantabria, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mayoral-van Son J, Juncal-Ruiz M, Ortiz-Garcia de la Foz V, Vazquez-Bourgon J, Setien-Suero E, Tordesillas-Gutierrez D, Gomez-Revuelta M, Ayesa-Arriola R, Crespo-Facorro B; PAFIP Research Group. Long-term clinical and functional outcome after antipsychotic discontinuation in early phases of non-affective psychosis: Results from the PAFIP-10 cohort. Schizophr Res. 2021 Jun;232:28-30. doi: 10.1016/j.schres.2021.04.011. Epub 2021 May 16. No abstract available. PMID 34004383